CLINICAL TRIAL: NCT01787188
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Fixed-Dose, Parallel-Group, Efficacy, and Safety Study of Meloxicam SoluMatrix™ Capsules in Patients With Pain Due to Osteoarthritis of the Knee or Hip
Brief Title: Study of Meloxicam Capsules to Treat Osteoarthritis Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEL3-12-02
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Meloxicam Test Capsules low dose QD (Experimental): Meloxicam Test Capsules low dose QD
  Interventions: Drug: Meloxicam Test Capsules
- Meloxicam Test Capsules high dose QD (Experimental): Meloxicam Test Capsules high dose QD
  Interventions: Drug: Meloxicam Test Capsules
- Placebo Capsule QD (Placebo Comparator): Placebo Capsule QD
  Interventions: Drug: Placebo Capsules

INTERVENTIONS:
Drug: Meloxicam Test Capsules
  Arms: Meloxicam Test Capsules low dose QD
Drug: Meloxicam Test Capsules
  Arms: Meloxicam Test Capsules high dose QD
Drug: Placebo Capsules
  Arms: Placebo Capsule QD

SUMMARY:
The purpose of this study is to determine whether Meloxicam [Test] Capsules are safe and effective for the treatment of osteoarthritis pain of the knee or hip.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Functional Class I-III OA of the hip or knee
* Chronic user of nonsteroidal anti-inflammatory drugs (NDAIDs) and/or acetaminophen for OA pain
* Discontinued all analgesic therapy at Screening
* For women of child-bearing potential: a woman who is not pregnant and not nursing, and who is practicing an acceptable method of birth control

Exclusion Criteria:

* History of allergic reaction or clinically significant intolerance to acetaminophen, aspirin, or any NSAIDs, including meloxicam
* Requires continuous use of opioid or opioid combination products to control OA pain of the knee or hip
* Clinically significant unstable cardiac, respiratory, neurological, immunological, hematological, or renal disease
* Significant difficulties swallowing capsules or unable to tolerate oral medication
* Previous participation in another clinical study of Meloxicam Capsules or received any investigational drug or device or investigational therapy within 30 days before Screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles P Andrews, MD, Principal Investigator — Diagnostics Research Group; Eddie Armas, MD, Principal Investigator — Well Pharma Medical Research Corporation; Matthew Barton, MD, Principal Investigator — Office of Matthew Barton, MD; David Bouda, MD, Principal Investigator — Heartland Clinical Research, Inc; John Champlin, MD, Principal Investigator — Medical Center; David Chen, MD, Principal Investigator — Beacon Clinical Research, LLC; Melanie Christina, MD, Principal Investigator — Clinical Investigations of Texas, LLC; James R Clark, MD, Principal Investigator — Charlottesville Medical Research Center, LLC; Stephen Daniels, DO, Principal Investigator — Premier Research Group - Austin; Richard R Eckert, MD, Principal Investigator — Hypothetest, LLC; Brandon Essink, MD, Principal Investigator — Meridian Clinical Research; John Flinchbaugh, DO, Principal Investigator — Fleming Island Center for Clinical Research; Neil Fraser, MD, Principal Investigator — Troy Internal Medicine, PC / Research Department; Richard M Glover, MD, Principal Investigator — Heartland Research Associates, LLC; John M Hill, MD, Principal Investigator — Avail Clinical Research; Curtis S Horn, MD, Principal Investigator — Quality Research Inc; Jeffry Jacqmein, MD, Principal Investigator — Jacksonville Center For Clinical Research; Richard Montgomery, MD, Principal Investigator — Triad Clinical Research; Alan Kivitz, MD, Principal Investigator — Altoona Center for Clinical Research; James Kopp, MD, Principal Investigator — Radiant Research, Inc; Gregory F Lakin, DO, Principal Investigator — Professional Research Network of Kansas, LLC; Sathish Modugu, MD, Principal Investigator — Drug Trials America; Julie Mullen, DO, Principal Investigator — Sterling Research Group, Ltd; Thomas Nussdorfer, MD, Principal Investigator — Medical Research Associates, Inc; Naynesh Patel, MD, Principal Investigator — Wells Institute for Health Awareness; Kashyap Patel, MD, Principal Investigator — Peninsula Research, Inc; Stephen J Poland, MD, Principal Investigator — Community Research; Larry D Reed, MD, PhD, Principal Investigator — Healthcare Research; Erich Schramm, MD, Principal Investigator — St. Johns Center for Clinical Research; Douglas R Schumacher, MD, Principal Investigator — Radiant Research, Inc; Louis Stephens, MD, Principal Investigator — Palmetto Clinical Trial Services, LLC; Mark Stich, DO, Principal Investigator — Westside Center for Clinical Research; Haydn M Thomas, MD, Principal Investigator — Clinical Trials Technology Inc; Susann Varano, MD, Principal Investigator — Clinical Research Consulting; Larkin T Wadsworth, MD, Principal Investigator — Sundance Clinical Research, LLC; Robert J Wagner, MD, Principal Investigator — Community Research; Matthew A Wenker, MD, Principal Investigator — Sterling Research Group, Ltd; Hayes T Williams, MD, PhD, Principal Investigator — Achieve Clinical Research, LLC; James Maynard, MD, Principal Investigator — Community Research; Roger Guthrie, MD, Principal Investigator — Arroyo Medical Group, Inc
Locations (39):
- United States (39):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Medical Center, Carmichael, California
  - Arroyo Medical Group, Inc, Pismo Beach, California
  - Clinical Research Consulting, Milford, Connecticut
  - Avail Clinical Research, DeLand, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Well Pharma Medical Research Corporation, Miami, Florida
  - Peninsula Research, Inc, Ormond Beach, Florida
  - St Johns Center for Clinical Research, Ponte Vedra, Florida
  - Heartland Research Associates, LLC, Newton, Kansas
  - Clinical Trials Technology Inc, Prairie Village, Kansas
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Community Research, Crestview Hills, Kentucky
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - Medical Research Associates, Inc, Traverse City, Michigan
  - Troy Internal Medicine, PC / Research Department, Troy, Michigan
  - Healthcare Research, Hazelwood, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Heartland Clinical Research, Inc, Omaha, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Office of Matthew Barton, MD, Las Vegas, Nevada
  - Drug Trials America, Hartsdale, New York
  - Triad Clinical Research, Greensboro, North Carolina
  - Sterling Research Group, Ltd, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Community Research - Anderson, Cincinnati, Ohio
  - Radiant Research, Inc, Columbus, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Radiant Research, Inc, Anderson, South Carolina
  - Palmetto Clinical Trial Services, LLC, Clinton, South Carolina
  - Premier Research - Austin, Austin, Texas
  - Clinical Investigations of Texas, LLC, Plano, Texas
  - Quality Research Inc, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Hypothetest, LLC, Roanoke, Virginia

REFERENCES:
- [Derived] Altman R, Hochberg M, Gibofsky A, Jaros M, Young C. Efficacy and safety of low-dose SoluMatrix meloxicam in the treatment of osteoarthritis pain: a 12-week, phase 3 study. Curr Med Res Opin. 2015 Dec;31(12):2331-43. doi: 10.1185/03007995.2015.1112772. PMID 26503347

RESULTS

PARTICIPANT FLOW:
Groups:
- Meloxicam 5 mg Once Daily: Meloxicam 5 mg: Capsules
- Meloxicam 10 mg Once Daily: Meloxicam 10 mg: Capsules
- Placebo: Placebo: Capsule
Period: Overall Study
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Started | 139 | 130 | 134
Completed | 122 | 112 | 116
Not Completed | 17 | 18 | 18
Not completed — Adverse Event | 2 | 4 | 6
Not completed — Lack of Efficacy | 7 | 3 | 5
Not completed — Non-compliance with Study Drug | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 2
Not completed — Protocol Violation | 3 | 2 | 3
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Other, including patient moved | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Subjects in this population received at least 1 dose of study drug and were analyzed according to treatment received, not treatment randomized. One subject who entered the study in the placebo group withdrew before receiving study drug. One subject who was randomized to meloxicam 5 mg received meloxicam 10 mg and was analyzed in that group
Groups:
- Total: Total of all reporting groups
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo | Total
Number analyzed (Participants) | 138 | 131 | 133 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.05) | 60.2 (8.77) | 61.1 (9.26) | 60.7 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 84 | 92 | 265
  Male | 49 | 47 | 41 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 11 | 33
  Not Hispanic or Latino | 128 | 119 | 122 | 369
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Subjects were allowed to select more than one race; therefore, some subjects are counted multiple times.
  participants
    American Indian or Alaska Native | 2 | 1 | 0 | 3
    Asian | 0 | 1 | 0 | 1
    Black or African-American | 27 | 29 | 23 | 79
    Native Hawaiian or Other Pacific Islander | 2 | 2 | 0 | 4
    White | 108 | 98 | 110 | 316
Weight [Mean (Standard Deviation); unit: kg] | 89.0 (17.00) | 85.9 (16.82) | 89.2 (17.27) | 88.1 (17.06)
Height [Mean (Standard Deviation); unit: cm] | 168.9 (10.28) | 167.9 (9.66) | 168.6 (10.37) | 168.5 (10.10)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (4.77) | 30.5 (5.31) | 31.3 (4.95) | 30.9 (5.01)
Baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score [Mean (Standard Deviation); unit: mm] — The pain in osteoarthritis subjects within the past 24 hours was measured at baseline using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score. The WOMAC pain subscale score is calculated as the mean of the visual analogue scale scores from 5 pain subscale questions, with 0 mm meaning "No Pain" and 100 mm meaning "Worst Possible Pain".
  The pain subscore was calculated for 139 subjects in the Meloxicam 5 mg group, 130 in the Meloxicam 10 mg group, and 133 in the placebo group.
  mm | 72.51 (15.360) | 72.19 (13.938) | 73.20 (15.472) | 72.64 (14.922)
Baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Function Subscore [Mean (Standard Deviation); unit: mm] — The function in osteoarthritis subjects within the past 24 hours was measured at baseline using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function subscale score. The WOMAC function subscale score is calculated as the mean of the visual analogue scale scores from 17 function subscale questions, with 0 mm meaning "No Functional Limitation" and 100 mm meaning "Worst Possible Functional Limitation".
  The function subscale score was calculated for 138 subjects in the Meloxicam 5 mg group, 130 in the Meloxicam 10 mg group, and 132 in the placebo group.
  mm | 66.83 (18.051) | 67.66 (16.873) | 68.61 (17.623) | 67.69 (17.505)
Baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscore [Mean (Standard Deviation); unit: mm] — The stiffness in osteoarthritis subjects within the past 24 hours was measured at baseline using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) stiffness subscale score. The WOMAC stiffness subscale score is calculated as the mean of the visual analogue scale scores from 2 stiffness subscale questions, with 0 mm meaning "No Stiffness" and 100 mm meaning "Worst Possible Stiffness".
  The stiffness subscale score was calculated for 139 subjects in the Meloxicam 5 mg group, 130 in the Meloxicam 10 mg group, and 132 in the placebo group.
  mm | 70.30 (18.367) | 69.19 (19.569) | 72.65 (17.056) | 70.71 (18.363)
Baseline Total Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score [Mean (Standard Deviation); unit: mm] — The pain, stiffness, and physical function in subjects with osteoarthritis were measured at baseline using the total Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scale. The total WOMAC score is the average of the mean visual analogue scale scores, with 0 mm meaning "No Limitation" and 100 mm meaning "Extreme Limitation".
  Baseline total WOMAC score was calculated for 138 subjects in the Meloxicam 5 mg once daily group, 130 subjects in the Meloxicam 10 mg once daily group, and 131 subjects in the placebo group.
  mm | 68.27 (16.315) | 68.74 (15.193) | 69.75 (16.134) | 68.91 (15.870)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 After Trial Entry in Osteoarthritis Pain Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score.
Description: The pain in subjects with osteoarthritis was measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score. The WOMAC pain subscale score is calculated as the average of the visual analogue scale (VAS) scores from 5 pain subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their pain level over the last 24 hours, with 0 mm representing "No Pain" and 100 mm representing "Extreme Pain".
  The WOMAC pain subscale score difference is calculated as the WOMAC pain subscale score assessed at Week 12 minus the WOMAC pain subscale score assessed at baseline.
Time Frame: Baseline to Week 12/Early Termination
Population: Intent-to-Treat Population. All subjects who received at least 1 dose of trial drug and had available measurements at the time specified.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 131 | 119 | 127
mm | -36.52 (2.485) | -34.41 (2.678) | -25.68 (2.636)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Difference in Least Squares Mean = -10.84, 95% CI 2-sided [-16.93 to -4.75], Standard Error of Mean 3.097
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0059, Mixed Models Analysis; Difference in Least Squares Mean = -8.74, 95% CI 2-sided [-14.94 to -2.53], Standard Error of Mean 3.154

2. Secondary Outcome: Change From Baseline to Week 2 After Trial Entry in Osteoarthritis Pain Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score.
Description: The pain in subjects with osteoarthritis was measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score. The WOMAC pain subscale score is calculated as the average of the visual analogue scale (VAS) scores from 5 pain subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their pain level over the last 24 hours, with 0 mm representing "No Pain" and 100 mm representing "Extreme Pain".
  The WOMAC pain subscale score difference was calculated as the WOMAC pain subscale score assessed at Week 2 minus the WOMAC pain subscale score assessed at baseline.
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 136 | 123 | 132
mm | -26.12 (2.217) | -20.42 (2.397) | -16.51 (2.367)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Difference in Least Squares Mean = -9.61, 95% CI 2-sided [-14.80 to -4.42], Standard Error of Mean 2.641
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.1486, Mixed Models Analysis; Difference in Least Squares Mean = -3.90, 95% CI 2-sided [-9.20 to 1.40], Standard Error of Mean 2.696

3. Secondary Outcome: Change From Baseline to Week 6 After Trial Entry in Osteoarthritis Pain Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score.
Description: The pain in subjects with osteoarthritis was measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score. The WOMAC pain subscale score is calculated as the average of the visual analogue scale (VAS) scores from 5 pain subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their pain level over the last 24 hours, with 0 mm representing "No Pain" and 100 mm representing "Extreme Pain".
  The WOMAC pain subscale score difference was calculated as the WOMAC pain subscale score assessed at Week 6 minus the WOMAC pain subscale score assessed at baseline.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 134 | 121 | 126
mm | -31.31 (2.339) | -30.82 (2.531) | -20.98 (2.503)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Difference in Least Squares Mean = -10.33, 95% CI 2-sided [-15.97 to -4.70], Standard Error of Mean 2.865
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Difference in Least Squares Mean = -9.84, 95% CI 2-sided [-15.58 to -4.10], Standard Error of Mean 2.917

4. Secondary Outcome: Change From Baseline to the Average of Weeks 2, 6, and 12 After Trial Entry in Osteoarthritis Pain Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score.
Description: The pain in subjects with osteoarthritis was measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score. The WOMAC pain subscale score is calculated as the average of the visual analogue scale (VAS) scores from 5 pain subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their pain level over the last 24 hours, with 0 mm representing "No Pain" and 100 mm representing "Extreme Pain".
  The WOMAC pain subscale score difference was calculated as the WOMAC pain subscale score assessed at Weeks 2, 6, and 12 minus the WOMAC pain subscale score assessed at baseline.
Time Frame: Baseline to Week 12/Early Termination
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 139 | 128 | 133
mm | -30.51 (2.151) | -27.89 (2.337) | -20.07 (2.318)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in Least Squares Mean = -10.44, 95% CI 2-sided [-15.40 to -5.48], Standard Error of Mean 2.521
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0024, ANCOVA; Difference in Least Squares Mean = -7.82, 95% CI 2-sided [-12.85 to -2.78], Standard Error of Mean 2.561

5. Secondary Outcome: Change From Baseline to Week 2 After Trial Entry in Osteoarthritis Pain, Stiffness, and Function Measured Using the Total Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score.
Description: Pain, stiffness, and function in subjects with osteoarthritis were measured using the Western Ontario and McMaster Universities (WOMAC) Index, which is a 24-item questionnaire. The total WOMAC score is calculated as the average of the mean visual analogue scale (VAS) scores from the questions in the pain, stiffness, and function subscales. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their response to each of the questions, with 0 mm representing "No Pain, Stiffness, or Difficulty" and 100 mm representing "Extreme Pain, Stiffness, and Difficulty".
  The total WOMAC score difference was calculated as the total WOMAC score assessed at Week 2 minus the total WOMAC score assessed at baseline.
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 132 | 123 | 130
mm | -21.62 (2.214) | -15.67 (2.384) | -11.28 (2.365)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Difference in Least Squares Mean = -10.34, 95% CI 2-sided [-15.49 to -5.18], Standard Error of Mean 2.623
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0997, Mixed Models Analysis; Difference in Least Squares Mean = -4.39, 95% CI 2-sided [-9.63 to 0.84], Standard Error of Mean 2.662

6. Secondary Outcome: Change From Baseline to Week 6 After Trial Entry in Osteoarthritis Pain, Stiffness, and Function Measured Using the Total Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score.
Description: Pain, stiffness, and function in subjects with osteoarthritis were measured using the Western Ontario and McMaster Universities (WOMAC) Index, which is a 24-item questionnaire. The total WOMAC score is calculated as the average of the mean visual analogue scale (VAS) scores from the questions in the pain, stiffness, and function subscales. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their response to each of the questions, with 0 mm representing "No Pain, Stiffness, or Difficulty" and 100 mm representing "Extreme Pain, Stiffness, and Difficulty".
  The total WOMAC score difference was calculated as the total WOMAC score assessed at Week 6 minus the total WOMAC score assessed at baseline.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 133 | 121 | 124
mm | -25.86 (2.367) | -25.45 (2.554) | -16.03 (2.537)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Difference in Least Squares Mean = -9.83, 95% CI 2-sided [-15.54 to -4.11], Standard Error of Mean 2.905
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; Difference in Least Squares Mean = -9.42, 95% CI 2-sided [-15.22 to -3.62], Standard Error of Mean 2.951

7. Secondary Outcome: Change From Baseline to Week 12 After Trial Entry in Osteoarthritis Pain, Stiffness, and Function Measured Using the Total Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score.
Description: Pain, stiffness, and function in subjects with osteoarthritis were measured using the Western Ontario and McMaster Universities (WOMAC) Index, which is a 24-item questionnaire. The total WOMAC score is calculated as the average of the mean visual analogue scale (VAS) scores from the questions in the pain, stiffness, and function subscales. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their response to each of the questions, with 0 mm representing "No Pain, Stiffness, or Difficulty" and 100 mm representing "Extreme Pain, Stiffness, and Difficulty".
  The total WOMAC score difference was calculated as the total WOMAC score assessed at Week 12/early termination minus the total WOMAC score assessed at baseline.
Time Frame: Baseline to Week 12/Early Termination
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 130 | 119 | 125
mm | -29.85 (2.518) | -29.71 (2.706) | -19.72 (2.678)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis; Difference in Least Squares Mean = -10.13, 95% CI 2-sided [-16.32 to -3.94], Standard Error of Mean 3.147
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; Difference in Least Squares Mean = -9.98, 95% CI 2-sided [-16.27 to -3.69], Standard Error of Mean 3.198

8. Secondary Outcome: Change From Baseline to the Average of Weeks 2, 6, and 12 After Trial Entry in Osteoarthritis Pain, Stiffness, and Function Measured Using the Total Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score.
Description: Pain, stiffness, and function in subjects with osteoarthritis were measured using the Western Ontario and McMaster Universities (WOMAC) Index, which is a 24-item questionnaire. The total (composite) WOMAC score is calculated as the average of the mean visual analogue scale (VAS) scores from the questions in the pain, stiffness, and function subscales. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their response to each of the questions, with 0 mm representing "No Pain, Stiffness, or Difficulty" and 100 mm representing "Extreme Pain, Stiffness, and Difficulty".
  The total WOMAC score difference was calculated as the total WOMAC score assessed at Weeks 2, 6, and 12 minus the total WOMAC score assessed at baseline.
Time Frame: Baseline to Week 12/Early Termination
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 138 | 128 | 131
mm | -25.15 (2.205) | -22.83 (2.389) | -14.67 (2.379)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in Least Squares Mean = -10.47, 95% CI 2-sided [-15.57 to -5.37], Standard Error of Mean 2.593
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0020, ANCOVA; Difference in Least Squares Mean = -8.16, 95% CI 2-sided [-13.33 to -2.99], Standard Error of Mean 2.627

9. Secondary Outcome: Change From Baseline to Week 2 After Trial Entry in Osteoarthritis Function Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Function Subscale Score.
Description: The function in osteoarthritis subjects within the past 24 hours was measured at baseline using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function subscale score. The WOMAC function subscale score is calculated as the mean of the visual analogue scale scores from 17 function subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their functional limitation level over the last 24 hours, with 0 mm meaning "No Functional Limitation" and 100 mm meaning "Extreme Functional Limitation".
  The WOMAC function subscale score difference was calculated as the WOMAC function subscale score assessed at Week 2 minus the WOMAC function subscale score assessed at baseline.
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 132 | 123 | 131
mm | -20.45 (2.270) | -14.41 (2.445) | -10.00 (2.423)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Difference in Least Squares Mean = -10.45, 95% CI 2-sided [-15.73 to -5.17], Standard Error of Mean 2.686
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.1065, Mixed Models Analysis; Difference in Least Squares Mean = -4.41, 95% CI 2-sided [-9.77 to 0.95], Standard Error of Mean 2.725

10. Secondary Outcome: Change From Baseline to Week 6 After Trial Entry in Osteoarthritis Function Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Function Subscale Score.
Description: The function in osteoarthritis subjects within the past 24 hours was measured at baseline using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function subscale score. The WOMAC function subscale score is calculated as the mean of the visual analogue scale scores from 17 function subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their functional limitation level over the last 24 hours, with 0 mm meaning "No Functional Limitation" and 100 mm meaning "Extreme Functional Limitation".
  The WOMAC function subscale score difference was calculated as the WOMAC function subscale score assessed at Week 6 minus the WOMAC function subscale score assessed at baseline.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 133 | 122 | 125
mm | -24.41 (2.419) | -24.38 (2.608) | -14.73 (2.590)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; Difference in Least Squares Mean = -9.68, 95% CI 2-sided [-15.50 to -3.85], Standard Error of Mean 2.961
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis; Difference in Least Squares Mean = -9.65, 95% CI 2-sided [-15.56 to -3.74], Standard Error of Mean 3.006

11. Secondary Outcome: Change From Baseline to Week 12 After Trial Entry in Osteoarthritis Function Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Function Subscale Score.
Description: The function in osteoarthritis subjects within the past 24 hours was measured at baseline using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function subscale score. The WOMAC function subscale score is calculated as the mean of the visual analogue scale scores from 17 function subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their functional limitation level over the last 24 hours, with 0 mm meaning "No Functional Limitation" and 100 mm meaning "Extreme Functional Limitation".
  The WOMAC function subscale score difference was calculated as the WOMAC function subscale score assessed at Week 12/early termination minus the WOMAC function subscale score assessed at baseline.
Time Frame: Baseline to Week 12/Early Termination
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 130 | 121 | 126
mm | -28.21 (2.566) | -28.40 (2.752) | -17.95 (2.724)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis; Difference in Least Squares Mean = -10.26, 95% CI 2-sided [-16.54 to -3.97], Standard Error of Mean 3.194
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis; Difference in Least Squares Mean = -10.45, 95% CI 2-sided [-16.82 to -4.08], Standard Error of Mean 3.240

12. Secondary Outcome: Change From Baseline to the Average of Weeks 2, 6, and 12 After Trial Entry in Osteoarthritis Function Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Function Subscale Score.
Description: The function in osteoarthritis subjects within the past 24 hours was measured at baseline using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function subscale score. The WOMAC function subscale score is calculated as the mean of the visual analogue scale scores from 17 function subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their functional limitation level over the last 24 hours, with 0 mm meaning "No Functional Limitation" and 100 mm meaning "Extreme Functional Limitation".
  The WOMAC function subscale score difference was calculated as the WOMAC function subscale score assessed at Weeks 2, 6, and 12 minus the WOMAC function subscale score assessed at baseline.
Time Frame: Baseline to Week 12/Early Termination
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 138 | 128 | 132
mm | -23.78 (2.254) | -21.70 (2.441) | -13.26 (2.429)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in Least Squares Mean = -10.52, 95% CI 2-sided [-15.72 to -5.31], Standard Error of Mean 2.646
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0018, ANCOVA; Difference in Least Squares Mean = -8.44, 95% CI 2-sided [-13.71 to -3.17], Standard Error of Mean 2.680

13. Secondary Outcome: Change From Baseline to Week 2 After Trial Entry in Osteoarthritis Stiffness Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score.
Description: The stiffness in osteoarthritis subjects within the past 24 hours was measured at baseline using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) stiffness subscale score. The WOMAC stiffness subscale score is calculated as the mean of the visual analogue scale scores from 2 stiffness subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their stiffness level over the last 24 hours, with 0 mm meaning "No Stiffness" and 100 mm meaning "Extreme Stiffness".
  The WOMAC stiffness subscale score difference was calculated as the WOMAC stiffness subscale score assessed at Week 2 minus the WOMAC stiffness subscale score assessed at baseline.
Time Frame: Baseline to Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 136 | 123 | 131
mm | -19.84 (2.381) | -14.88 (2.578) | -8.86 (2.545)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Difference in Least Squares Mean = -10.98, 95% CI 2-sided [-16.55 to -5.41], Standard Error of Mean 2.831
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0379, Mixed Models Analysis; Difference in Least Squares Mean = -6.02, 95% CI 2-sided [-11.71 to -0.34], Standard Error of Mean 2.890

14. Secondary Outcome: Change From Baseline to Week 6 After Trial Entry in Osteoarthritis Stiffness Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score.
Description: The stiffness in osteoarthritis subjects within the past 24 hours was measured at baseline using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) stiffness subscale score. The WOMAC stiffness subscale score is calculated as the mean of the visual analogue scale scores from 2 stiffness subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their stiffness level over the last 24 hours, with 0 mm meaning "No Stiffness" and 100 mm meaning "Extreme Stiffness".
  The WOMAC stiffness subscale score difference was calculated as the WOMAC stiffness subscale score assessed at Week 6 minus the WOMAC stiffness subscale score assessed at baseline.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 134 | 121 | 125
mm | -26.52 (2.559) | -23.39 (2.767) | -14.30 (2.737)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Difference in Least Squares Mean = -12.22, 95% CI 2-sided [-18.42 to -6.02], Standard Error of Mean 3.152
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0049, Mixed Models Analysis; Difference in Least Squares Mean = -9.10, 95% CI 2-sided [-15.41 to -2.78], Standard Error of Mean 3.210

15. Secondary Outcome: Change From Baseline to Week 12 After Trial Entry in Osteoarthritis Stiffness Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score.
Description: The stiffness in osteoarthritis subjects within the past 24 hours was measured at baseline using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) stiffness subscale score. The WOMAC stiffness subscale score is calculated as the mean of the visual analogue scale scores from 2 stiffness subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their stiffness level over the last 24 hours, with 0 mm meaning "No Stiffness" and 100 mm meaning "Extreme Stiffness".
  The WOMAC stiffness subscale score difference was calculated as the WOMAC stiffness subscale score assessed at Week 12/early termination minus the WOMAC stiffness subscale score assessed at baseline.
Time Frame: Baseline to Week 12/Early Termination
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 131 | 119 | 126
mm | -29.68 (2.691) | -28.10 (2.902) | -18.74 (2.857)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; Difference in Least Squares Mean = -10.94, 95% CI 2-sided [-17.55 to -4.33], Standard Error of Mean 3.359
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0066, Mixed Models Analysis; Difference in Least Squares Mean = -9.36, 95% CI 2-sided [-16.09 to -2.63], Standard Error of Mean 3.422

16. Secondary Outcome: Change From Baseline to the Average of Weeks 2, 6, and 12 After Trial Entry in Osteoarthritis Stiffness Measured on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score.
Description: The stiffness in osteoarthritis subjects within the past 24 hours was measured at baseline using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) stiffness subscale score. The WOMAC stiffness subscale score is calculated as the mean of the visual analogue scale scores from 2 stiffness subscale questions. Subjects mark the VAS, which is a horizontal line 100 mm in length, with a single vertical line to indicate their stiffness level over the last 24 hours, with 0 mm meaning "No Stiffness" and 100 mm meaning "Extreme Stiffness".
  The WOMAC stiffness subscale score difference was calculated as the WOMAC stiffness subscale score assessed at Weeks 2, 6, and 12 minus the WOMAC stiffness subscale score assessed at baseline.
Time Frame: Baseline to Week 12/Early Termination
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Number analyzed (Participants) | 138 | 128 | 132
mm | -24.76 (2.345) | -21.33 (2.548) | -13.09 (2.526)
Statistical Analysis 1: Comparison: Meloxicam 5 mg Once Daily vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in Least Squares Mean = -11.67, 95% CI 2-sided [-17.08 to -6.26], Standard Error of Mean 2.751
Statistical Analysis 2: Comparison: Meloxicam 10 mg Once Daily vs Placebo; Test type: Superiority or Other; p = 0.0034, ANCOVA; Difference in Least Squares Mean = -8.24, 95% CI 2-sided [-13.74 to -2.74], Standard Error of Mean 2.795

ADVERSE EVENTS:
Description: Subjects in this population received at least 1 dose of study drug and were analyzed according to treatment received, not treatment randomized. One subject who entered the study in the placebo group withdrew before receiving study drug. One subject who was randomized to meloxicam 5 mg received meloxicam 10 mg and was analyzed in that group
Arm/Group | Meloxicam 5 mg Once Daily | Meloxicam 10 mg Once Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 0/138 | 0/131 | 0/133
Other Adverse Events (participants affected / at risk) | 14/138 | 13/131 | 10/133
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Meloxicam 5 mg Once Daily (N=138) | Meloxicam 10 mg Once Daily (N=131) | Placebo (N=133)
Diarrhea (Gastrointestinal disorders) | 4 | 3 | 1
Headache (Nervous system disorders) | 2 | 5 | 4
Nausea (Gastrointestinal disorders) | 3 | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3
Urinary Tract Infection (Infections and infestations) | 3 | 2 | 3
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No